CLINICAL TRIAL: NCT05722340
Title: Video-assisted Thoracic Surgery for Lung Biopsy Using Non-intubated (NIVATS) Versus Intubated General Anaesthesia (IGAVATS): a Randomized, Controlled, Pilot Trial Addressing Biopsy Quality in Undetermined Interstitial Lung Diseases
Brief Title: NIVATS Versus IGAVATS: a Pilot Trial Addressing Biopsy Quality in Undetermined Interstitial Lung Diseases
Acronym: NIVATS-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Grace Asso (Groupe francophone de Réhabilitation Améliorée après Chirurgie) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RECHMPL 22_0042
Record Dates: First submitted 2023-01-18; First posted 2023-02-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: In this prospective, parallel group, randomized (1:1), controlled, pilot trial, screening will take place during routine multidisciplinary assessment (MDA) meetings. The study is then presented to eligible patients during their next pre-surgical visits; if the patients are interested in participating, informed consent procedures are completed (again during routine visits) and the patients are randomized to two arms. In the experimental arm, patients will undergo NIVATS for lung biopsy, and in the standard arm, patients will undergo traditional IGAVATS for lung biopsy. Histology is then performed as usual, before entering a centralized pathway for a second analysis by an expert external to the study, and a second routine MDA convened (both blinded to study arms). Patients are followed-up for 12 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To assure the blinding of non-surgical study staff (MDA participants, histologists, etc), allocation results in the electronic case report (eCRF) form are made available to designated surgical staff only. Patients, investigators / outcome assessors / care givers and study staff are blinded to allocation results in as much as possible.
  Only designated surgical staff (identified prior to centre initiation and kept to a strict necessary minimum) not otherwise involved in outcome assessment or patient care have access to allocation results on the eCRF and are summoned to maintain secrecy.
  Data analysts will not be involved in trial field logistics and will be blinded. During analyses, when group assignments are first required, they will only be revealed as "group A" or "group B". Only when analyses have been completed will the exact nature of groups be revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIVATS (Experimental): Lung biopsy is performed using non-intubated video-assisted thoracic surgery (NIVATS).
  Interventions: Procedure: Non-intubated video-assisted thoracic surgery (NIVATS) for lung biopsy
- IGAVATS (Active Comparator): Lung biopsy is performed using Intubated general anaesthesia video-assisted thoracic surgery (IGAVATS).
  Interventions: Procedure: Intubated general anaesthesia video-assisted thoracic surgery (IGAVATS) for lung biopsy

INTERVENTIONS:
Procedure: Non-intubated video-assisted thoracic surgery (NIVATS) for lung biopsy — An epidural anaesthesia associated with mild sedation requiring no ventilation is used.
  Arms: NIVATS
Procedure: Intubated general anaesthesia video-assisted thoracic surgery (IGAVATS) for lung biopsy — Uses a traditional deep anaesthesia and one-lung ventilation
  Arms: IGAVATS

SUMMARY:
The main objective of this study is to compare two independent groups of patients requiring lung biopsy for undetermined interstitial lung disease (ILD) in terms of diagnostic confidence as determined by histologists.

DETAILED DESCRIPTION:
The primary objective of this study is to compare two independent groups of patients requiring lung biopsy for undetermined interstitial lung disease (ILD) in terms of diagnostic confidence as determined by histologists. The experimental arm will be operated under a neoteric non-intubated video assisted thoracic surgery (NIVATS) technique and the comparator arm under a usual intubated general anaesthesia video-assisted thoracic surgery (IGAVATS) technique.

Secondarily, the two groups will also be compared in terms of: (i) further variables associated with histology, biopsy quality and size; (ii) surgical performance, (iii) patient trajectories and lung function; (iv) quality of life, and (v) harms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with purported interstitial lung disease
* Patient requiring a surgical lung biopsy to reinforce diagnosis according to current recommendations and validated by a multidisciplinary assessment
* Minimum age: 18 years

Exclusion Criteria:

* Contra-indication for surgery
* Uncontrolled oesophageal gastric reflux despite optimal treatment
* Thoracic deformation (For example, pectus excavatum/carinatum or major scoliosis)
* Risk of pleural adhesion (For example, patient who has already undergone thoracic surgery)
* History of abnormal bleeding
* Predictable risk of difficult intubation
* Body mass index (BMI) > 30
* Severe cardiovascular comorbidity (For example, instable ischemic cardiomyopathy)
* Unable to comply with all trial procedures/visits (For example, language barriers, upcoming move of household to another region, unwillingness to schedule the required followup visits.)
* Protected populations according to the French Public Health Code Articles L1121-5,6,8 (For example, pregnant, parturient or lactating women, prisoners, adults under guardianship or otherwise unable to consent.)
* Potential interference from another study (The patient is participating in another interventional study, or has done so in the past month, or is affected by an exclusion period stipulated by a previous study.)
* Non-beneficiary of the French single-payer national medical insurance system
* Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-11-24 (Estimated)

PRIMARY OUTCOMES:
The level of diagnostic confidence based on centralized histology only | Day 1 to day 15
  The level of diagnostic confidence for a given diagnosis is established according to a quantitative scale ranging from '0' (absolute rule-out) to '10' (diagnostic certainty). A visual guide for scale use is provided with scores <1 corresponding to "alternate diagnosis", scores >=1 and <4 corresponding to "indeterminate", scores >=4 and <7 corresponding to "probable", and scores >=7 corresponding to "highly probable" categories.

SECONDARY OUTCOMES:
The level of diagnostic confidence based on routine histology only | Day 1 to day 15
  The level of diagnostic confidence for a given diagnosis is established according to a quantitative scale ranging from '0' (absolute rule-out) to '10' (diagnostic certainty). A visual guide for scale use is provided with scores <1 corresponding to "alternate diagnosis", scores >=1 and <4 corresponding to "indeterminate", scores >=4 and <7 corresponding to "probable", and scores >=7 corresponding to "highly probable" categories.
The level of diagnostic confidence achieved at multidisciplinary assessment (MDA)-2 | Day 7 to day 28
  The level of diagnostic confidence for a given diagnosis is established according to a quantitative scale ranging from '0' (absolute rule-out) to '10' (diagnostic certainty). A visual guide for scale use is provided with scores <1 corresponding to "alternate diagnosis", scores >=1 and <4 corresponding to "indeterminate", scores >=4 and <7 corresponding to "probable", and scores >=7 corresponding to "highly probable" categories.
Change in the level of diagnostic confidence for the most favoured diagnosis between multidisciplinary assessment (MDA)-1 and multidisciplinary assessment (MDA)-2 | Day 7 to day 28
  The level of diagnostic confidence for a given diagnosis is established according to a quantitative scale ranging from '0' (absolute rule-out) to '10' (diagnostic certainty). A visual guide for scale use is provided with scores <1 corresponding to "alternate diagnosis", scores >=1 and <4 corresponding to "indeterminate", scores >=4 and <7 corresponding to "probable", and scores >=7 corresponding to "highly probable" categories.
Classification according to ATS/ERS at MDA-1 | Day -28 to day -3
  Classification according to the American Thoracic Society / European Respiratory society: Alternative diagnosis / Indeterminate / Probable / Highly probable
Classification according to ATS/ERS at MDA-2 | Day 7 to day 28
  Classification according to the American Thoracic Society / European Respiratory society: Alternative diagnosis / Indeterminate / Probable / Highly probable
Inter-histologist concordance for ATS/ERS categories | Day 1 to 15
  Inter-histologist concordance for ATS/ERS categories
Longest length (mm) of biopsy specimens | Day 1 to 15
  Longest length (mm) of biopsy specimens
Volume (cc) of biopsy specimens | Day 1 to 15
  Volume (cc) of biopsy specimens
Weight (g) of biopsy specimens | Day 1 to 15
  Weight (g) of biopsy specimens
Numerical scale for biopsy quality | Day 1 to 15
  The histologist ranks biopsy quality from worst imaginable (0) to excellent (10).
Preparation time (minutes) | Day 0
  Minutes lapsed between entering the surgical ward and entering the operating room (OR)
OR time (minutes) | Day 0
  Minutes lapsed between entering and exiting the OR
Recovery room (RR) time (minutes) | Day 0
  Minutes lapsed between exiting the OR and exiting the surgical ward.
Post-RR time (hours) | Day 1 to 15
  Hours lapsed between exit from surgical ward, and discharge from hospital
First drink time (minutes) | Day 0
  Minutes lapsed between application of last bandage on surgical wounds to first drink
Post-operative fasting time (hours) | Day 0
  Hours lapsed between application of last bandage on surgical wounds to first meal
Time with chest tube in place (hours) | Day 0
  Hours lapsed between application of last bandage on surgical wounds to removal of chest tube
Visual analogue scale score for post-operative pain | Day 1, morning after surgery
  The patient will be asked to evaluate his/her level of post-operative pain using a numeric rating scale (0-10) the morning after surgery where 0 represents no pain, and 10 represents the worse possible pain.
Patient satisfaction (satisfied vs unsatisfied) | Hospital discharge (expected maximum of 15 days)
  The patient will be asked to evaluate his/her satisfaction (satisfied vs unsatisfied)
Time to dischargeability | Days 1 to 15
  Dischargeability is defined as meeting the following criteria: (i) satisfactory pain control via oral analgesia; (ii) ability to mobilize and return to usual autonomy; (iii) absence of clinical, laboratory and radiological complications; (iv) stable respiratory state compatible pre-surgical state and home discharge; (v) vital signs are normal for the patient; (vi) chest tube removal >12 hours.
Length of initial hospitalization stay (hours) | Expected maximum of 15 days
  Length of initial hospitalization stay (hours)
Cumulative days of hospitalization | 12 months
  Cumulative days of hospitalization
Cumulative days of exacerbation | 12 months
  Cumulative days of exacerbation
Days alive, not exacerbating and not in hospital | 12 months
  Days alive, not exacerbating and not in hospital
Forced vital capacity (litres) | Day -28 to Day -1
  Forced vital capacity (litres)
Forced vital capacity (litres) | 12 months
  Forced vital capacity (litres)
Forced vital capacity (% theoretical value) | Day -28 to Day -1
  Forced vital capacity (% theoretical value)
Forced vital capacity (% theoretical value) | 12 months
  Forced vital capacity (% theoretical value)
Euroqol 5 dimensions 5 levels questionnaire: mobility dimension score | Day -28 to Day -1
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: mobility dimension score | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: self-care dimension score | Day -28 to Day -1
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: self-care dimension score | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: usual activities dimension score | Day -28 to Day -1
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: usual activities dimension score | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: pain/discomfort dimension score | Day -28 to Day -1
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: pain/discomfort dimension score | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: anxiety/depression dimension score | Day -28 to Day -1
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Euroqol 5 dimensions 5 levels questionnaire: anxiety/depression dimension score | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
Presence / absence of complications | 12 months
  Complications will be listed and classified (Minor: (1) Any complication without need for pharmacologic treatment or other intervention; (2) Any complication that requires pharmacologic treatment or minor intervention only; Major: (3) Any complication that requires surgical, radiologic, endoscopic intervention, or multitherapy; (3a) Intervention does not require general anesthesia; (3b) Intervention requires general anesthesia; (4) Any complication requiring intensive care unit management and life support; (4a) Single organ dysfunction; (4b) Multiorgan dysfunction; (5) Any complication leading to the death of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'Anesthésie et Réanimation Cardiothoracique - CHU Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study.
  Data will be made available to persons who address a reasonable request to the study director.
  Individual participant data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  The study protocol, participant Information materials, worksheet and data sharing plan will also be made available to the public.
Supporting Information: Study Protocol, ICF
Time Frame: Datasets that underlie the results reported in the article (text, tables, figures, and appendices) can be requested after the publication process has been completed.
  The study protocol will be published in an open-access, peer-reviewed journal. Other key documents will be made available on the Open Science Framework as they are finalized.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * If the data do not fulfil the requirements of the reference methodology (MR-00X) (ex: data about religion, etc.), the appropriate CNIL approval has to be obtained by the user.
  * If the data will be used outside the European Union, standard contractual clauses have to be signed between Montpellier University Hospital and the user before sharing data.
URL: https://osf.io/dnbfg/